CLINICAL TRIAL: NCT03003065
Title: Safety and Tumoricidal Effect of Low Dose Temoporfin Photodynamic Therapy in Patients With Inoperable Bile Duct Cancers (Foscan® Study)
Brief Title: Safety and Tumoricidal Effect of Low Dose Foscan PDT in Patients With Inoperable Bile Duct Cancers
Acronym: PDT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Foscan
Record Dates: First submitted 2016-02-24; First posted 2016-12-26 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cholangiocarcinoma; Tumor; Klatskin Tumor
Keywords: Inoperable cholangiocarcinoma; Photodynamic therapy; Endoscopic retrograde cholangiopancreatography
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasms; Klatskin Tumor | interventions — temoporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Foscan (Other): A single treatment with Temoporfin (Foscan) 3 mg given intravenously followed by PDT with laser light at 652 nm (Ceralas, Biolitec, Germany) within 72 hours
  Interventions: Drug: Temoporfin

INTERVENTIONS:
Drug: Temoporfin — A single treatment with Temoporfin (Foscan) 3 mg given intravenously followed by PDT with laser light at 652 nm (Ceralas, Biolitec, Germany) within 72 hours
  Other Names: Foscan

SUMMARY:
In this study, we hope to evaluate the safety of PDT using temoporfin plus endoscopic stents in patients with inoperable bile duct cancers. In addition as a preliminary study we sought to determine if the treatment can reduce tumor volume in the short term.

DETAILED DESCRIPTION:
Cholangiocarcinoma is a tumor associated with a grave prognosis. The only curative treatment is surgery or liver transplantation. Only about 10-20% of patients with the tumor are operated upon. In the majority of patients, the tumor is often diagnosed at a late stage. Many patients are not operated upon owing to their advanced age or comorbid illnesses. These patients suffer from intense pruritus a result of obstructive jaundice, recurrent biliary sepsis and progressive hepatic failure leading to death. Quality in life in these patients is poor. The median survival in these patients is around 6 months. The palliative treatment is stents inserted either at ERCP or through a percutaneous transhepatic route. Many return with recurrent cholangitis necessitating frequent stent changes. Photodynamic therapy (PDT) in combination with stenting is the only proven treatment that confers a survival benefit when compared to stenting alone. Two randomized controlled trials have shown significant survival advantage in patients treated by PDT in addition to stenting compared to stenting alone. Ortner et al. 1 randomized 39 patients with inoperable cholangiocarinoma to endoscopic stents with or without PDT. Median survival in those given PDT was 493 days compared to that of 98 days in those with stents alone. Survival difference was again wide in favor of PDT use in another randomized controlled study by Zoepf et al 2 (median survival 630 vs. 210 days). In addition, PDT improves quality of life and cholestasis in patients with cholangiocarcinoma. In a series from Germany, survival after PDT and stenting compared favorably to R1 and R2 resections. 3 Despite of the evidence, PDT for inoperable cholangiocarcinoma is not available in Hong Kong.

Meso-tetrahydroxyphenylchlorin (mTHPC, Foscan®) is a photosensitizer for PDT in cholangiocarcinoma. In compared with other agents such as Photofin and Photosan, PDT treatment using temoporfin at a low dose (3 mg per treatment) is associated with a deeper tissue penetration (4-6mm) and a reduced period of photosensitivity.

In this study, we hope to evaluate the safety of PDT using temoporfin plus endoscopic stents in patients with inoperable bile duct cancers. In addition as a preliminary study we sought to determine if the treatment can reduce tumor volume in the short term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable cholangiocarcinoma belonging to all Bismuth Corlette classification.
* Karnofsky index >30%
* Satisfactory relief of jaundice (serum bilirubin < 100µmol/L) with biliary prostheses inserted either at ERCP or via percutaneous transhepatic routes.
* Absence of biliary sepsis
* Age 18-80
* Provision of written consent
* No evidence of metastatic disease

Exclusion Criteria:

* Porphyria
* Previous inserted metallic biliary stents
* Refusal to provide a written consent.
* Moribund from disseminated disease or comorbidities
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Safety (will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0) | 10 years
  Safety (will be graded according to the Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
Tumor response as categorized by the World Health Organization criteria at 8 weeks as assessed by ERCP and Intraduct ultrasound | 10 years
  Tumor response as categorized by the World Health Organization criteria at 8
Relief of jaundice at 8 weeks (<50% pretreatment serum bilirubin) | 10 years
  Relief of jaundice at 8 weeks (<50% pretreatment serum bilirubin)
Cholangitis and stent occlusions requiring stent change (will be assessed based on blood tests and ERCP findings) | 10 years
  Cholangitis and stent occlusions requiring stent change (will be assessed based on blood tests and ERCP findings)
Quality of life (in every visit, European Organization for Research and Treatment of Cancer core questionnaire [EORTC QLQ-C30] will be filled and specific symptom enquiry is made; itchiness, fever and general well-being over a Likert 0-4 scale. | 10 years
  Quality of life (in every visit, European Organization for Research and Treatment of Cancer core questionnaire [EORTC QLQ-C30] will be filled and specific symptom enquiry is made; itchiness, fever and general well-being over a Likert 0-4 scale.

CONTACTS AND LOCATIONS:
Overall Officials: James YW LAU, MD, Principal Investigator — CUHK
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No